CLINICAL TRIAL: NCT02798614
Title: A Comparison of Radiographic and Clinical Results After Short Versus Conventional Plaster Cast Fixation Time in Reduced Distal Radius Fractures
Brief Title: Short Versus Conventional Plaster Cast Fixation Time in Reduced Distal Radius Fractures
Acronym: GitRa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Albert Christersson, MD, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GR-0102
Record Dates: First submitted 2016-06-01; First posted 2016-06-14 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Colles' Fracture
MeSH Terms: conditions — Colles' Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10-day cast (Active Comparator): Removal of plaster cast 10 Days after reduction
  Interventions: Device: 10-day cast
- 1-month cast (No Intervention): Removal of plaster cast 1 month after reduction

INTERVENTIONS:
Device: 10-day cast — Removal of plaster cast fixation 10 days after reduction
  Arms: 10-day cast

SUMMARY:
The purpose of this study is to compare the radiographic and clinical outcomes after short versus conventional plaster cast fixation time in reduced distal radius fractures.

DETAILED DESCRIPTION:
Displaced distal radius fractures treated with closed reduction and plaster cast fixation are radiographed 10 days (range 8-13 days) after reduction and randomized to one of two study arms; immediate removal of plaster cast or continued fixation in plaster cast for another 3 weeks. Radiographic and Clinical outcome measurements at 1, 4 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Distal radius fracture with intact ulna (except for processus styloideus ulnae)
* Dorsal angulation 5-40 degrees
* Axial compression < 4 mm
* Intra articular step-off < 1 mm
* Low energy trauma
* Closed fracture
* Suitable for treatment with closed reduction and plaster cast fixation

Exclusion Criteria:

* Fracture older than 3 Days
* Previously fractured ipsi- or contralateral wrist
* Dementia
* Inflammatory joint disorder

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2002-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Radiographic displacement | At admission, 10 days, 1 month and 12 months
  Change in dorsal angulation, radial angulation and axial compression between follow-ups.

SECONDARY OUTCOMES:
Grip strength | Uninjured side. Injured side at 1, 4 , 12 months
  Grip strength compared to uninjured side at 1, 4 and 12 months
Range of motion | Uninjured side. Injured side at 1, 4 and 12 months
  Range of motion in dorsal extension, volar flexion, supination and pronation compared to uninjured side at 1, 4 and 12 months.
Assessment of pain intensity | 10 days, 1, 4 and 12 months
  Average pain over the last 24 h assessed with a visual analogue scale (VAS) at 10 days, 1, 4 and 12 months
Assessment of functional outcome with three different functional assessment scores; 1,The modified de Bruijn wrist score 2, The modified Mayo wrist scoring chart 3, The Gartland and Werley Demerit wrist point system modified by Sarmiento. | 12 months
  The three functional assessment scores are composite outcome measures consisting of multiple measures (results to be reported as single values for each Group),

CONTACTS AND LOCATIONS:
Overall Officials: Albert Christersson, MD, Principal Investigator — Department of Orthopaedics, University Hospital of Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christersson A, Larsson S, Ostlund B, Sanden B. Radiographic results after plaster cast fixation for 10 days versus 1 month in reduced distal radius fractures: a prospective randomised study. J Orthop Surg Res. 2016 Nov 21;11(1):145. doi: 10.1186/s13018-016-0478-7. PMID 27871284